CLINICAL TRIAL: NCT02150798
Title: The Effects of a High Fat and Low Carbohydrate Diet on Clinical Status in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, LILIA CASTILLO MARTINEz, at the National Institute of Medical Science and Nutrition Salvador Zubiran, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIC001
Record Dates: First submitted 2014-05-09; First posted 2014-05-30 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Diet Therapy; Diet, Carbohydrate Restricted; Fatty Acids, Omega 3; Oximetry; phase angle; Triglycerides, blood; Lipids, blood; Hand Strength; Body Composition; Electric Impedance
MeSH Terms: conditions — Heart Failure | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat and low carbohydrate diet (Experimental): High fat low carbohydrate diet composition was 40 % of carbohydrates, 40 % of lipids (12 % saturated, 18 % monounsaturated and 10% polyunsaturated, ) and 20 % of protein for two months
  Interventions: Other: High fat and low carbohydrate diet
- Control diet (Active Comparator): the standard diet composition was 50 % of carbohydrates, 30 % of lipids (10 % saturated, 10 % polyunsaturated, and 10 % monounsaturated) and 20 % of protein for two months
  Interventions: Other: Control diet

INTERVENTIONS:
Other: High fat and low carbohydrate diet — high fat and low carbohydrate diet. At baseline and at 2 month of following, the variables that were evaluated,
  Arms: High fat and low carbohydrate diet
Other: Control diet — Control diet. At baseline and at 2 month of following, the variables that were evaluated,
  Arms: Control diet

SUMMARY:
The aim of the present study was to evaluate the effects of a high fat, low carbohydrate (CHO) diet on clinical status during 60 days of follow-up in patients with stable heart failure (HF).

In a randomized controlled clinical trial 44 ambulatory patients with HF were included, assigned to an intervention (40% CHO, 40% fat and 20% protein; n=22) or control groups (50% CHO, 30% fat, 20% protein; n=20). Both groups received recommended pharmacological management. At baseline and at 2 months of follow-up, the variables evaluated were: body composition, handgrip strength, oxygen saturation, dietary intake, clinical data, lipid profile, plasma glucose and exercise tolerance

DETAILED DESCRIPTION:
Nutritional therapy in patients with heart failure (HF) has been focused on fluid and sodium restriction to decrease volume overload. This has proved to decrease extracellular water levels, which manifests as a reduction in edema. Also, in patients with HF and preserved ejection fraction, reduction of sodium in addition to the Dietary Approaches to Stop Hypertension (DASH) diet has been associated with improved left ventricular diastolic function and arterial elasticity, reduced blood pressure, and modestly lower mortality in HF women.

Some studies focused on reducing cardiovascular risk suggest that saturated fatty acids should be replaced by some other macronutrient. Clinical trials which evaluated the replacement of saturated fatty acids with monounsaturated or polyunsaturated fatty acids have found an improvement in blood lipid concentrations and reduced cardiovascular risk in different populations. In the case of omega (n)-3 polyunsaturated fatty acids (PUFA), antiarrhythmic, antithrombotic, anti-atherogenic, and anti-inflammatory effects , improvement of endothelial function, lower blood pressure and plasma triglycerides, and reduced mortality and admission to the hospital for cardiovascular reasons have been documented in patients with chronic heart failure. In addition, the Mediterranean diet, which is high in monounsaturated fatty acids, was associated with cardiovascular risk reduction in other populations.

In HF PUFA was associated with better systolic and diastolic function, but with no effect on mortality. On the other hand, the replacement of saturated fatty acids by carbohydrates must be considered responsible for the possible increase in total cholesterol, LDL cholesterol (LDL-c), plasma triglycerides and decreased HDL cholesterol. Furthermore, the metabolism of carbohydrates induces higher oxygen consumption (VO2), higher carbon dioxide (VCO2) production and increased minute ventilation (VE). In other populations, it has been associated with lower respiratory efficiency and decreased exercise tolerance.

HF should be considered a complex condition in which the heart fails to deliver enough oxygen-rich blood to meet the body's needs, and these patients characteristically have skeletal muscle dysfunction and compromised pulmonary function and ventilatory response, with peak oxygen consumption reduced and deterioration of their clinical state.

Nonetheless, nutritional therapy of HF patients has not been focused on optimizing mechanical ventilation with improved consumption of oxygen. Moreover, studies that examine nutritional therapy in HF have not evaluated the ventilatory response. Therefore, we propose to evaluate the effects of a high fat and low carbohydrate diet on clinical status of chronic stable HF patients.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of heart failure
* New York Heart Association functional classes I to III

Exclusion Criteria:

* New Year Heart Association functional classes IV symptoms
* Patients with severe renal insufficiency (estimated glomerular filtration rate <30 mL/min per 1.73 m2) - Patients with hepatic failure
* Patients with specific dietary regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | 2 months after intervention
  Oxygen saturation was measured indirectly with a pulse oximeter

SECONDARY OUTCOMES:
Handgrip strength | 2 months after intervention
  Handgrip strength was evaluated with a dinamometer
Blood pressure | 2 months after intervention
  Blood pressure was evaluated with an automatic sphygmomanometer
Exercise tolerance | 2 months after intervention
  Exercise tolerance was measured in metabolic equivalents (METs) with symptom-limited treadmill exercise testing, conducted according to the modified Bruce protocol
Adverse effects | 2 months follow-up
  Symptoms such as constipation, abdominal distension, nausea or diarrhea were evaluated

OTHER OUTCOMES:
Body composition | 2 month after intervention
  Bioimpedance parameters: resistance, reactance, phase angle, body water

CONTACTS AND LOCATIONS:
Overall Officials: Dulce G Gonzalez, M.Sc., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Lilia Castillo, M.Sc., Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Arturo Orea, MD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Gabriela Olvera, B.Sc, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Karla Balderas, B.Sc., Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Cira Santillán, M.Sc., Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Wendy Rodríguez, M.Sc., Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico